CLINICAL TRIAL: NCT02864927
Title: Postmarketing Surveillance Study for Use of Meningococcal (Groups A, C, Y and W-135) Polysaccharide Diphtheria Toxoid Conjugate Vaccine (Menactra®) in the Republic of Korea
Brief Title: Postmarketing Surveillance Study for Use of Menactra® in the Republic of Korea
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MTA79; U1111-1174-4708 (Other: WHO)
Record Dates: First submitted 2016-08-05; First posted 2016-08-12 (Estimated); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Meningitis; Meningococcal Meningitis; Meningococcal Infections
Keywords: Meningitis; Meningococcal Meningitis; Meningococcal Infections; Menactra®; Meningococcal Vaccine
MeSH Terms: conditions — Meningitis; Meningitis, Meningococcal; Meningococcal Infections | interventions — Meningococcal Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Menactra Group 1 (Experimental): Participants aged 9 to 23 months will receive 2 doses of Menactra
  Interventions: Biological: Meningococcal (Groups A, C, Y and W 135) Polysaccharide Diphtheria Toxoid Conjugate Vaccine
- Menactra Group 2 (Experimental): Participants aged 2 to 55 years will receive 1 dose of Menactra
  Interventions: Biological: Meningococcal (Groups A, C, Y and W 135) Polysaccharide Diphtheria Toxoid Conjugate Vaccine

INTERVENTIONS:
Biological: Meningococcal (Groups A, C, Y and W 135) Polysaccharide Diphtheria Toxoid Conjugate Vaccine — 0.5 mL, Intramuscular. 2 doses 3 months apart
  Other Names: Menactra®
  Arms: Menactra Group 1
Biological: Meningococcal (Groups A, C, Y and W 135) Polysaccharide Diphtheria Toxoid Conjugate Vaccine — 0.5 mL, Intramuscular
  Other Names: Menactra®
  Arms: Menactra Group 2

SUMMARY:
The purpose of the study is to perform the re-examination of Menactra® administered in the routine clinical settings in accordance with the Ministry of Food and Drug Safety regulation.

Primary objective:

* To describe the safety profile after 1 dose of Menactra® administered from 9 months to 55 years of age under standard health care practice.

DETAILED DESCRIPTION:
Subjects aged 9 months through 55 years and who are given study vaccine during routine health-care visits will be enrolled in the study.

They will be followed-up for up to Day 42 following vaccination.

No study vaccine will be supplied or administered as part of this study, subjects will be monitored following routine vaccine administration in clinical settings.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent form signed by the subject (for subjects from 19 to 55 years of age) or the parent(s) or other legal representative (for subjects from 9 months to 18 years of age)
* Receipt of one dose of Menactra® (on the day of inclusion) according to approved local product insert paper .

Exclusion Criteria:

* Participation at the time of study enrollment (or in the 4 weeks preceding the study vaccination) or planned participation during the present study period in another clinical study investigating a vaccine, drug, medical device, or a medical procedure
* Subjects who already participated in this study.

Ages: 9 Months to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1311 (Actual)
Dates: Start 2016-07-21 (Actual); Primary Completion 2019-06-12 (Actual); Study Completion 2019-06-12 (Actual)

PRIMARY OUTCOMES:
Number of Participants Reporting Solicited Injection-Site Reactions and Systemic Reactions Following Vaccination with Menactra® | Day 0 up to Day 30 post-vaccination
  Solicited injection-site reactions: Tenderness/Pain, Erythema, and Swelling. Solicited systemic reactions: infants and toddlers (9 to 23 months) Fever (temperature), Vomiting, Abnormal crying, Drowsiness, Loss of appetite and Irritability; Subjects aged 2 to 55 years, Fever (temperature), Headache, Malaise, and Myalgia
Number of Participants Reporting Unsolicited Adverse Events Following Vaccination with Menactra® | Day 0 up to Day 30 post-vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi Pasteur, a Sanofi Company
Locations (1):
- Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Kim HS, Engel S, Neveu D, Thollot Y, Oster P, Yang K. Post-Marketing Surveillance Observational Study of Quadrivalent Meningococcal Diphtheria Toxoid Conjugate Vaccine (MenACWY-DT, MCV4/Menactra(R)) in the Republic of Korea, 2014-2019. Infect Dis Ther. 2021 Mar;10(1):399-409. doi: 10.1007/s40121-020-00393-4. Epub 2021 Jan 13. PMID 33439463